CLINICAL TRIAL: NCT00675584
Title: Childhood Asthma Research and Education (CARE) Network Trial - Maintenance Versus Intermittent Inhaled Steroids in Wheezing Toddlers (MIST)
Brief Title: CARE Network Maintenance Versus Intermittent Inhaled Steroids in Wheezing Toddlers (MIST)
Acronym: MIST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Vernon M. Chinchilli, PhD, Professor and Chair, Department of Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 581; 5U10HL064313 (NIH); 5U10HL064288 (NIH); 5U10HL064305 (NIH); 5U10HL064295 (NIH); 5U10HL064287 (NIH); 5U10HL064307 (NIH)
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Results first posted 2012-06-01 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Budesonide (Active Comparator): Participants will receive 0.5 mg of ICS (budesonide as Pulmicort Respules®) once a day at night, except during respiratory tract illnesses. During respiratory tract illnesses, participants will receive placebo each morning and 0.5 mg of budesonide each night for 7 days.
  Interventions: Drug: Budesonide; Drug: Placebo Budesonide
- Budesonide (Experimental): Participants will receive 1 mg of ICS (budesonide as Pulmicort Respules®) twice a day for 7 days at the onset of a respiratory tract illness; they will receive placebo ICS once a day at all other times during the study.
  Interventions: Drug: Budesonide; Drug: Placebo Budesonide

INTERVENTIONS:
Drug: Budesonide — Participants in Arm 1 will receive 0.5 mg of budesonide once a day. Participants in Arm 2 will receive 1 mg of budesonide twice a day for 7 days at the onset of respiratory tract illnesses.
  Other Names: Pulmicort Respules®
Drug: Placebo Budesonide — Participants in Arm 1 will receive placebo budesonide each morning during respiratory tract illnesses for 7 days. Participants in Arm 2 will receive placebo budesonide once a day for the entire study, other than when they have a respiratory tract illness.
  Other Names: Placebo Pulmicort Respules®

SUMMARY:
Asthma affects about 4 million children in the United States and is a leading cause of hospitalizations and school absenteeism. Continuous wheezing in very young children may develop into asthma. Low doses of inhaled corticosteroids (ICS) are commonly prescribed to treat children with particularly bad wheezing episodes. This study will compare the safety and effectiveness of low doses of ICS taken daily versus higher doses of ICS taken only during respiratory tract illnesses for toddlers with continuous wheezing or coughing illnesses.

DETAILED DESCRIPTION:
Childhood asthma can be caused by many factors, including allergens, cigarette smoke, air pollution, or infections. Symptoms include wheezing, shortness of breath, chest tightness, and coughing. Wheezing illnesses are common during the first several years of life, and continuous wheezing, or recurrent intermittent wheezing, may be an indicator of asthma. Recurrent intermittent wheezing can also lead to breathing difficulties, sleep disturbances, and severe exacerbations that result in emergency department visits, hospitalizations, or even death. The Prevention of Early Asthma in Kids (PEAK) and Acute Intervention Management Strategies (AIMS) studies, both of which are part of the Childhood Asthma Research and Education (CARE) Network, as well as several other studies, have identified therapies that may improve recurrent wheezing in young children. This study will compare the safety and effectiveness of two treatment regimens-low doses of ICS taken on a daily basis versus higher doses of ICS taken only during respiratory tract illnesses-at improving recurrent wheezing in toddlers. Study researchers will also identify individual characteristics (e.g., age, gender, family history of asthma and allergies, the degree of allergy, genetics) that may be associated with treatment response. Lastly, the relationship of virus infections to respiratory illnesses, wheezing episodes, and response to study treatments will also be studied.

This study will enroll children between 12 and 53 months of age who have experienced episodes of wheezing or coughing in the year before study entry, with at least one episode that required one of the following: oral steroids, an urgent unscheduled medical visit, an emergency room visit, or hospitalization. This study will begin with a 2-week evaluation period during which potential participants will receive placebo once a day. Parents will document their child's asthma symptoms and medication use in a daily diary. Next, at a baseline study visit, eligible participants will be randomly assigned to one of the following two 12-month treatment groups:

* Group 1 participants will receive a low dose of ICS once a day at night, except during respiratory tract illnesses. During a respiratory tract illness, participants will receive placebo each morning and a low dose of ICS each night for 7 days.
* Group 2 participants will receive a high dose of ICS twice a day for 7 days during each respiratory illness and placebo once a day at night at all other times.

Throughout the 12 months of treatment, all participants will receive albuterol to treat respiratory symptoms and prednisolone if asthma symptoms worsen. Parents will be given an action plan to help manage their child's symptoms, and during respiratory illnesses, parents will contact study researchers to determine the best treatment plan. Study visits will occur at baseline and Weeks 4, 12, 20, 28, 36, 44, and 52. Participants' parents will take part in scheduled telephone interviews one month after each clinic visit to provide information on their child's asthma symptoms, study medication use, and health problems. Most study visits will include a physical exam and lung function testing. At select study visits, the following will occur: allergy skin testing, blood collection, nasal mucus sampling, and parent questionnaires to assess asthma, quality of life, and environmental factors. A portion of the participants' blood will undergo genetic analysis; a blood collection from parents for genetic analysis will be optional. Throughout the treatment period, participants' parents will record asthma symptoms and medication usage in a daily diary.

ELIGIBILITY:
Inclusion Criteria at Screening Visit:

Participants who meet all of the following criteria are eligible for study entry. Participants may be reassessed if not initially eligible.

* Positive asthma predictive index (API) status
* A history of at least 4 wheezing episodes in the prior year with at least one physician diagnosed or at least 3 wheezing episodes in the prior year with at least one physician diagnosed and at least 3 months of asthma controller therapy in the prior year
* Experienced a severe exacerbation requiring systemic corticosteroids, urgent unscheduled or emergency visit, or hospitalization in the 12 months before the screening visit
* All immunizations must be completed, including varicella (unless the child has already had clinical varicella). If the child needs the varicella vaccine, this will be arranged with the primary care physician and must be received before study entry.
* Allows blood to be used for genetic analysis
* Willingness to provide informed consent by the child's parent or guardian

Exclusion Criteria at Screening Visit:

Participants who meet any of the following criteria are NOT eligible for enrollment, but they may be re-enrolled if these exclusion criteria disappear:

* Use of more than six courses of systemic corticosteroids in the 12 months before the screening visit
* More than two hospitalizations for wheezing illnesses in the 12 months before the screening visit
* Use of oral or systemic corticosteroids in the 2 weeks before the screening visit
* Current treatment with antibiotics for diagnosed sinus disease
* Current participation or has participated in the month before the screening visit in another investigational drug trial
* Evidence that the family may be unreliable or nonadherent, or may move from the clinical center area before trial completion
* Medically unable to use systemic corticosteroids
* Clinically relevant gastroesophageal reflux
* Inability of the child to cooperate with nebulizer therapy

Participants who meet any of the following criteria are NOT eligible for enrollment, and they may not be re-enrolled:

* Gestation less than late preterm, as defined as birth before 34 weeks gestational age
* Significant developmental delay/failure to thrive, defined as crossing of two major percentile lines during the last year for age and gender. If a child plots less than the 10th percentile for age and gender, a growth chart for the previous year will be obtained from the child's primary care provider.
* Head circumference less than the 3rd percentile or greater than the 97th percentile unless medical evaluation documents no associated illness
* Presence of lung disease other than asthma, such as cystic fibrosis and bronchopulmonary dysplasia (BPD). Evaluation during the screening process will assure that an adequate evaluation of other lung diseases has been performed.
* Presence of other significant medical illnesses (e.g., cardiac, liver, gastrointestinal, endocrine) that would place the child at increased risk of participating in the study
* Immunodeficiency disorders
* History of respiratory failure requiring mechanical ventilation
* History of hypoxic seizure
* History of significant adverse reaction to any study medication ingredient

Exclusion Criteria at Baseline Visit:

Participants will be ineligible to continue in the study and be randomly assigned to a treatment group if any of the following is documented during the 2-week observation period, but they may be re-enrolled if these exclusion criteria disappear:

* Persistent symptomatic asthma, as defined as experiencing symptoms requiring albuterol use on average three or more days per week or two or more night time awakenings due to asthma-associated symptoms
* Inadequate adherence (less than 75% of days) to diary card completion or nebulizer medication use
* Use of any asthma medication except albuterol (used on as needed basis)

Ages: 12 Months to 53 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 278 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David T. Mauger, PhD, Principal Investigator — Penn State College of Medicine; Stanley J. Szefler, MD, PhD, Principal Investigator — National Jewish Health; Robert F. Lemanske, Jr., MD, Principal Investigator — University of Wisconsin, Madison; Robert S. Zeiger, MD, PhD, Principal Investigator — Kaiser Permanente Medical Center; Robert C. Strunk, MD, Principal Investigator — Washington University School of Medicine; Fernando D. Martinez, MD, Principal Investigator — University of Arizona College of Medicine; Lynn M. Taussig, MD, Study Chair — University of Denver
Locations (5):
- United States (5):
  - University of Arizona College of Medicine, Tucson, Arizona
  - Kaiser Permanente Medical Center, San Diego, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Washington University School of Medicine, St Louis, Missouri
  - University of Wisconsin - Madison, Madison, Wisconsin

REFERENCES:
- [Result] Zeiger RS, Mauger D, Bacharier LB, Guilbert TW, Martinez FD, Lemanske RF Jr, Strunk RC, Covar R, Szefler SJ, Boehmer S, Jackson DJ, Sorkness CA, Gern JE, Kelly HW, Friedman NJ, Mellon MH, Schatz M, Morgan WJ, Chinchilli VM, Raissy HH, Bade E, Malka-Rais J, Beigelman A, Taussig LM; CARE Network of the National Heart, Lung, and Blood Institute. Daily or intermittent budesonide in preschool children with recurrent wheezing. N Engl J Med. 2011 Nov 24;365(21):1990-2001. doi: 10.1056/NEJMoa1104647. PMID 22111718
- See also: Click here for the Childhood Asthma Research and Education (CARE) Network Web site — http://www.asthma-carenet.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Daily Budesonide: Participants will receive 0.5 mg of ICS (budesonide as Pulmicort Respules®) once a day at night, except during respiratory tract illnesses. During respiratory tract illnesses, participants will receive placebo each morning and 0.5 mg of budesonide each night for 7 days.
- Intermittent Budesonide: Participants will receive 1 mg of ICS (budesonide as Pulmicort Respules®) twice a day for 7 days at the onset of a respiratory tract illness; they will receive placebo ICS once a day at all other times during the study.
Period: Overall Study
Arm/Group | Daily Budesonide | Intermittent Budesonide
Started | 139 | 139
Completed | 100 | 113
Not Completed | 39 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Budesonide | Intermittent Budesonide | Total
Number analyzed (Participants) | 139 | 139 | 278
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 139 | 139 | 278
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.9 (0.9) | 2.9 (0.9) | 2.9 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 37 | 86
  Male | 90 | 102 | 192
Region of Enrollment [Number; unit: participants]
  United States | 139 | 139 | 278

OUTCOME MEASURES:

1. Primary Outcome: Rate of Exacerbations Requiring Systemic Corticosteroids
Description: The rate of exacerbations was calculated as the number of exacerbations requiring prednisone per years of follow-up
Time Frame: Measured during the 12-month follow-up period
Population: Even if a child terminated prior to completion of the 12 months of follow-up, he/she contributed to the numerator and denominator of the exacerbation rate
Measure: Mean (95% Confidence Interval); unit: events per years of follow-up
Arm/Group | Daily Budesonide | Intermittent Budesonide
Number analyzed (Participants) | 139 | 139
events per years of follow-up | 0.97 [0.76 to 1.22] | 0.95 [0.75 to 1.20]

2. Secondary Outcome: Proportion of Episode-free Days
Description: An episode-free day consisted of no asthma symptoms and no asthma rescue medications
Time Frame: Measured during the 12-month follow-up period
Population: Even if a child terminated prior to completion of the 12 months of follow-up, he/she contributed to the numerator and denominator of the proportion of episode-free days
Measure: Mean (95% Confidence Interval); unit: proportion of episode-free days
Arm/Group | Daily Budesonide | Intermittent Budesonide
Number analyzed (Participants) | 139 | 139
proportion of episode-free days | 0.78 [0.76 to 0.81] | 0.78 [0.75 to 0.80]

3. Secondary Outcome: Number of Urgent Care Visits, Emergency Department Visits, or Hospitalizations for Wheezing or Asthma Per 12 Months
Time Frame: Measured during the 12-month follow-up period
Population: Even if a child terminated prior to completion of the 12 months of follow-up, he/she contributed to the number of urgent care visits
Measure: Mean (95% Confidence Interval); unit: visits per 12 months
Arm/Group | Daily Budesonide | Intermittent Budesonide
Number analyzed (Participants) | 139 | 139
visits per 12 months | 2.40 [1.91 to 3.02] | 2.37 [1.89 to 2.97]

4. Secondary Outcome: Number of Participants With Treatment Failure
Description: Treatment failure was defined as the occurrence of at least one of the following events:
  1. four courses of systemic corticosteroids
  2. one hospitalization for acute exacerbation of wheezing
  3. hypoxic seizure during an acute exacerbation of asthma/wheezing
  4. intubation for acute asthma/wheezing
  5. serious adverse event related to a study medication
  6. physician discretion with specific rationale
Time Frame: Measured during the 12-month follow-up period
Population: Even if a child terminated prior to completion of the 12 months of follow-up, his/her data were included in the assessment of treatment failure
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Budesonide | Intermittent Budesonide
Number analyzed (Participants) | 139 | 139
Participants | 17 | 9

5. Secondary Outcome: Change Between 12 Months and Baseline in Exhaled Nitric Oxide (eNO)
Description: Exhaled nitric oxide (eNO) is measured in parts per billion, and the change constructed between 12 months and baseline
Time Frame: baseline and 12 months
Population: Even if a child terminated prior to completion of the 12 months of follow-up, his/her data were included in the analysis based on the linear mixed-effects model
Measure: Least Squares Mean (95% Confidence Interval); unit: parts per billion
Arm/Group | Daily Budesonide | Intermittent Budesonide
Number analyzed (Participants) | 139 | 139
parts per billion | -0.14 [-0.32 to 0.04] | -0.18 [-0.38 to 0.02]

6. Secondary Outcome: Change Between 12 Months and Baseline in Pulmonary Reactance and Resistance Measured Via Oscillometry
Time Frame: baseline and 12 months
Population: Prior to enrollment of the first randomized study participant, the clinical investigators decided that it would be futile to perform oscillometry in children of the target age range for MIST (2-5 years of age). A previous CARE Network trial (PEAK) performed oscillometry in such children, but the data were highly variable and of poor quality.
Arm/Group | Daily Budesonide | Intermittent Budesonide
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Adverse Events Associated With Corticosteroid Use
Time Frame: Measured during the 12-month follow-up period
Population: All randomized children are included
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Budesonide | Intermittent Budesonide
Number analyzed (Participants) | 139 | 139
Participants | 3 | 0

8. Secondary Outcome: Number of Days of Absence From Daycare and Preschool for the Child and From Work for the Caregiver Per 12 Months
Time Frame: Measured during the 12-month follow-up period
Population: Even if a child terminated prior to completion of the 12 months of follow-up, he/she contributed to the number of days
Measure: Mean (95% Confidence Interval); unit: days per 12 months
Arm/Group | Daily Budesonide | Intermittent Budesonide
Number analyzed (Participants) | 139 | 139
days per 12 months | 3.02 [2.22 to 4.12] | 2.72 [2.00 to 3.70]

9. Secondary Outcome: Proportion of Days With Rescue Albuterol Use
Time Frame: Measured during the 12-month follow-up period
Population: Even if a child terminated prior to completion of the 12 months of follow-up, he/she contributed to the number of days
Measure: Mean (95% Confidence Interval); unit: proportion of days
Arm/Group | Daily Budesonide | Intermittent Budesonide
Number analyzed (Participants) | 139 | 139
proportion of days | 0.05 [0.04 to 0.06] | 0.06 [0.05 to 0.07]

10. Secondary Outcome: Change in Wheeze Severity During a Respiratory Tract Illness
Description: Wheeze severity is scored as 0 (none) to 5 (very severe) during a respiratory tract illness
Time Frame: Measured during the first seven days for each respiratory tract illness
Population: The data from every respiratory tract illness is included in the analysis
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Daily Budesonide | Intermittent Budesonide
Number analyzed (Participants) | 139 | 139
units on a scale | 0.5 [0.1 to 0.8] | 0.8 [0.5 to 1.1]

11. Secondary Outcome: Change Between 12 Months and Baseline in the Caregiver Quality-of-life
Description: The caregiver quality-of-life questionnaire consists of seven questions, each scored from 0 (worse) to 3 (best), and all seven questions are summed to yield a total score ranging from 0 to 21
Time Frame: baseline and 12 months
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Daily Budesonide | Intermittent Budesonide
Number analyzed (Participants) | 139 | 139
units on a scale | 1.4 [-3.0 to 5.8] | 2.0 [-1.8 to 5.8]

ADVERSE EVENTS:
Time Frame: 1 year
Description: does not differ from the clinicaltrials.gov definitions
Arm/Group | Daily Budesonide | Intermittent Budesonide
Serious Adverse Events (participants affected / at risk) | 7/139 | 10/139
Other Adverse Events (participants affected / at risk) | 9/139 | 11/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Budesonide (N=139) | Intermittent Budesonide (N=139)
hospitalization due to exacerbation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
other (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Budesonide (N=139) | Intermittent Budesonide (N=139)
nausea or vomiting (Gastrointestinal disorders) | 9 (9) | 11 (11)

LIMITATIONS AND CAVEATS:
May not be applicable to young children whose asthma is more severe than that of the children in the study. Daily or intermittent use of inhaled glucocorticoids may not be efficacious in preschool-age children with transient or infrequent wheezing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No